CLINICAL TRIAL: NCT04094168
Title: Clinical Outcomes of Del Nido Cardioplegia in Adult Cardiac Surgery: a Randomized Controlled Trial
Brief Title: Clinical Impact of Del Nido Cardioplegia in Adult Cardiac Surgery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: JESSICA GARCIA SUAREZ (Other)
Responsible Party: Sponsor-Investigator, JESSICA GARCIA SUAREZ, Principal investigator, Puerta de Hierro University Hospital
Organization: Puerta de Hierro University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: EUDRA CT 2017-005144-14
Record Dates: First submitted 2019-09-13; First posted 2019-09-18 (Actual); Last update posted 2025-07-22 (Actual); Status verified 2025-07

CONDITIONS: Heart; Surgery, Heart, Functional Disturbance as Result
Keywords: Del Nido Cardioplegia; Cardioplegia; Adult Cardiac Surgery; Myocardial protection; Heart surgery
MeSH Terms: interventions — Del Nido cardioplegia solution

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Del Nido Cardioplegia solution (Experimental): 1 liter of Del Nido cardioplegia after aortic cross-clamp will be given. Additional dose will be applied if aortic cross-clamp exceeds 90 minutes or whenever cardiac activity is observed.
  Interventions: Drug: DEL NIDO CARDIOPLEGIA
- Cold blood Cardioplegia solution (Active Comparator): Administering of cardioplegia using current standard of care blood-based cardioplegia protocol. An induction dose of whole blood cardioplegia will be given at a temperature of 4-8 degrees, with subsequent doses of cardioplegia every 20 minutes or whenever cardiac activity is observed.
  Interventions: Drug: COLD BLOOD BASED CARDIOPLEGIA

INTERVENTIONS:
Drug: DEL NIDO CARDIOPLEGIA — Del Nido components: Plasmalyte 148 (1000 ml), NaHCO3 8.4% 1M (13 ml), MgSO4 0,5 M (16,5 ml), Mannitol 20% (16,3 ml), KCl 2 M (13 ml), Lidocaine 2% (6,5 ml).
  Electrolytic composition (l000 ml): Na+ 153 mEq, K+ 31 mEq, Cl - 124 mEq, Mg2+ 19,5 mEq, NaHCO3 13 mEq, Acetate 27 mEq, Sulfate 16,5 mEq, Gluconate 23 mEq.
  Arms: Del Nido Cardioplegia solution
Drug: COLD BLOOD BASED CARDIOPLEGIA — Cardibraun components: Electrolytic composition (1000 ml): Na+ 185,8 mmol, K+ 24,1 mmol, Cl- 192,8 mmol, Acetate 23 mmol, Fosfate 0,97 mmol, Citrate 6,32 mmol.
  Other Names: CARDIBRAUN
  Arms: Cold blood Cardioplegia solution

SUMMARY:
Cardioplegia solutions have been used for myocardial protection in cardiac surgery for decades. Different cardioplegic strategies have been evaluated.

Del Nido cardioplegia was initially used in pediatric patients and has been expanding into adult cardiac centers over the last decade. It can be used as a single dose and it is a reasonable tool do decrease cardioplegic interventions. Recent meta-analysis based on 9 retrospective studies has shown that "clinical outcomes of Del Nido cardioplegia are noninferior to the outcomes of conventional cardioplegia in adult cardiac surgery".

To assess the potencial benefits of Del Nido cardioplegia we performed this clinical trial to evaluate superiority of Del Nido cardioplegia compared to cold blood cardioplegia in terms of myocardial protection and clinical-related outcomes. 474 participants will be randomized either into Del Nido cardioplegia protocol or into the cold blood cardioplegia protocol. Perioperative outcomes will be presented.

DETAILED DESCRIPTION:
This clinical trial is performed at Puerta de Hierro Hospital in Spain. The protocol has been approved by institutional ethical committee and Spanish Agency of medicines and medical devices (AEMPS).

The aim of the study is to evaluate superiority of Del Nido cardioplegia solution compared to cold blood cardioplegia solution in terms of myocardial protection and clinical-related outcomes.

According to results in recent meta-analysis, the author estimated a total sample size of 474 participants to give 80 % of power at the 5% significant level.

Participants aged 18 years or older undergoing elective cardiac surgery are randomized 1:1 to receive Del Nido cardioplegia solution (study group) and cold blood cardioplegia solution (control group).

Primary outcome will be assessed by biochemical variables of myocardial injury (troponin T level at inmediate post-op, 3-12 hours, 12-24 hours, 24-48 hours post-op); and clinical variables: "Presence of acute myocardial infarction within 72 hours after surgery", "Prolonged low cardiac output", "Prolonged postoperative vasoplegia" within 48 hours after surgery and/or "Ventricular tachyarrythmias" within 24 hours after surgery.

Secondary outcomes include intraoperative variables of myocardial protection (incidence of ventricular fibrillation, inotropic and vasopressor support at the end of surgical intervention, cardiopulmonary bypass time, aortic cross-clamp time) and postoperative clinical outcomes variables (mechanical ventilation time, incidence of delirium, stroke, acute renal failure, atrial fibrillation, length of stay in intensive care unit, length of stay in hospital and In-hospital mortality).

ELIGIBILITY:
Inclusion Criteria:

* Patients age 18 years or older undergoing adult cardiac surgery.
* Elective surgical procedures requiring cardiopulmonary bypass and myocardial arrest.

Exclusion Criteria:

* Emergency surgery.
* Patients on preoperative inotropic support and/or mechanical circulatory support.
* Patient who refuse to participate in the study.
* Lidocaine allergy.
* Port access mitral valve surgery.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 474 (Actual)
Dates: Start 2018-06-15 (Actual); Primary Completion 2019-12-15 (Actual); Study Completion 2020-02-28 (Actual)

PRIMARY OUTCOMES:
Blood troponin levels. | Up to 48 hours
  Biochemical variables of myocardial injury: Blood troponin levels measured at admission in intensive care unit, 12, 24, 48 hours post-op.
Acute cardiovascular event. | Up to 72 hours
  Composite outcome of clinical events "Prolonged low cardiac output", "Prolonged postoperative vasoplegia", "Ventricular tachyarrythmias" and/or "Acute myocardial infarction".
  * Prolonged low cardiac output. Inotropic pharmacologic support more than 48 hours in intensive care unit and/or mechanical circulatory support.
  * Prolonged postoperative vasoplegia. Vasopressor support more than 48 hours in intensive care unit.
  * Ventricular tachyarrythmias. Ventricular fibrillation and hemodynamically unstable ventricular tachycardia within 24 hours after surgery.
  * Acute myocardial infarction within 72 hours after surgery.

SECONDARY OUTCOMES:
Ventricular fibrillation after aortic cross-clamp removal. | Intraoperative.
  Incidence of ventricular fibrillation after aortic cross-clamp removal (Y/N).
Defibrillation requirement. | Intraoperative.
  Defibrillation requirement after aortic cross-clamp removal (Y/N).
Cardioplegia delivery. | Intraoperative.
  Cardioplegia delivery (antegrade, retrograde, both).
Cardiopulmonary bypass time (CBP). | Intraoperative.
  Duration of cardiopulmonary bypass (CBP) (min).
Aortic cross-clamp time | Intraoperative.
  Duration of aortic cross-clamp time (min).
Return to cardiopulmonary bypass. | Intraoperative
  Failure to separate from cardiopulmonary bypass (Y/N).
Intraoperative packed red blood cells transfusion. | Intraoperative
  Intraoperative packed red blood cells transfusion (U).
Intraoperative maximal blood glucose concentration. | Intraoperative
  Intraoperative maximal blood glucose concentration (mg/dl).
Postoperative atrial fibrillation. | Up to 2 weeks.
  New-onset atrial fibrillation or hemodynamically unstable atrial fibrillation that requires treatment (Y/N).
Reoperation. | Up to 24 hours.
  Reoperation within 24 hours after surgery (Y/N).
Inotropic or vasopressor support in intensive care unit. | At admission in intensive care unit, 24, 48 hours.
  Inotropic or vasopressor support in intensive care unit (Y/N).
Duration of inotropic support after cardiopulmonary bypass. | Up to 2 weeks.
  Duration of inotropic support after cardiopulmonary bypass (hours).
Time to extubation. | Up to 2 weeks.
  Mechanical ventilation time (min).
Acute renal failure. | Up to 2 weeks.
  Incidence of renal failure (Requirement for postoperative renal replacement therapy) (Y/N).
Ischemic stroke. | Up to 2 weeks.
  Incidence of ischemic stroke (Y/N).
Delirium. | Up to 2 weeks.
  Incidence of delirium (Y/N).
Postoperative packed red blood cells transfusion. | Up to 1 week.
  Postoperative packed red blood cells transfusion (U)
Length of stay in intensive care unit | through study completion, an average 1 month.
  Length of stay in intensive care unit (days).
Length of stay in hospital | through study completion, an average 6 months.
  Length of stay in hospital (days).
Postoperative ventricular ejection fraction change. | through study completion, an average 6 months.
  Postoperative ventricular ejection fraction (LVEF) change (Y/N).
Mortality. | through study completion, an average 6 months.
  Mortality (Y/N).

CONTACTS AND LOCATIONS:
Locations (1):
- Puerta de Hierro Hospital, Majadahonda, Madrid, Spain

IPD SHARING:
Plan to Share IPD: Yes
All IPD that underlie results in a publication.
Supporting Information: Study Protocol, CSR
Time Frame: 6 months after publication.
Access Criteria: Access by mail to principal investigator: Jessica.suarez@gmail.com Access by mail to sponsor: apforteza@yahoo.es

REFERENCES:
- [Background] Buckberg GD, Athanasuleas CL. Cardioplegia: solutions or strategies? Eur J Cardiothorac Surg. 2016 Nov;50(5):787-791. doi: 10.1093/ejcts/ezw228. Epub 2016 Jul 1. No abstract available. PMID 27369117
- [Background] Ad N, Holmes SD, Massimiano PS, Rongione AJ, Fornaresio LM, Fitzgerald D. The use of del Nido cardioplegia in adult cardiac surgery: A prospective randomized trial. J Thorac Cardiovasc Surg. 2018 Mar;155(3):1011-1018. doi: 10.1016/j.jtcvs.2017.09.146. Epub 2017 Nov 13. PMID 29246552
- [Background] Li Y, Lin H, Zhao Y, Li Z, Liu D, Wu X, Ji B, Gao B. Del Nido Cardioplegia for Myocardial Protection in Adult Cardiac Surgery: A Systematic Review and Meta-Analysis. ASAIO J. 2018 May/Jun;64(3):360-367. doi: 10.1097/MAT.0000000000000652. PMID 28863040
- [Background] Lazar HL. del Nido cardioplegia: Passing fad or here to stay? J Thorac Cardiovasc Surg. 2018 Mar;155(3):1009-1010. doi: 10.1016/j.jtcvs.2017.09.126. Epub 2017 Oct 10. No abstract available. PMID 29110949
- [Background] Tam DY, Fremes SE. Del Nido cardioplegia: A one stop shot for adult cardiac surgery? J Thorac Cardiovasc Surg. 2018 Mar;155(3):1019-1020. doi: 10.1016/j.jtcvs.2017.10.066. Epub 2017 Oct 31. No abstract available. PMID 29198802
- [Derived] Garcia-Suarez J, Garcia-Fernandez J, Martinez Lopez D, Reques L, Sanz S, Carballo D, Martin CE, Ospina VM, Villar S, Martin A, Casado M, Villafranca A, Gonzalez AI, Serrano S, Forteza A. Clinical impact of del Nido cardioplegia in adult cardiac surgery: A prospective randomized trial. J Thorac Cardiovasc Surg. 2023 Nov;166(5):1458-1467. doi: 10.1016/j.jtcvs.2022.01.044. Epub 2022 Feb 8. PMID 35279289
- [Derived] Garcia-Suarez J, Garcia Fernandez J, Sanz S, Martinez Lopez D, Reques L, Forteza Gil A. Del Nido Cardioplegia Versus Cold Blood Cardioplegia in Adult Cardiac Surgery: Protocol for a Randomized Controlled Trial. JMIR Res Protoc. 2020 Jul 14;9(7):e17826. doi: 10.2196/17826. PMID 32673265